CLINICAL TRIAL: NCT00788905
Title: Uremic Toxin Removal, Blood Cell Kinetics, and Inflammatory Response in Patients Treated With the Allient System
Brief Title: Comparison of Conventional Dialysis and the Allient System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Renal Research Institute (Other)
Collaborators: Renal Solutions, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 065-08
Record Dates: First submitted 2008-09-23; First posted 2008-11-11 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: End Stage Renal Disease; Chronic Kidney Failure
Keywords: Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Subject will continue conventional hemodialysis therapy for one week ("no intervention" phase) and then swtich to the Allient system for two weeks ("active comparator" phase).
  Interventions: Device: Allient System

INTERVENTIONS:
Device: Allient System — The Allient System uses a different type of blood pump and a lower volume of dialysate.

SUMMARY:
The purpose of the study to determine whether the level of inflammation may be decreased, the lifespan of red blood cells increased and the clearance of waste products in the blood improved through the use of the Allient System as compared to conventional hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Maintenance in-center hemodialysis
* Age greater than or equal to 18 years
* Has been on hemodialysis for at least 4 months
* Uses a standard single-pass dialysis machine with a high-flux dialyzer

Exclusion Criteria:

* Hospitalization during the 8 weeks preceding enrollment
* Infection requiring antibiotic treatment during the 8 weeks preceding enrollment
* Central venous cather as dialysis access
* Uncontrollable blood coagulation anomalies
* Smokers
* Dialysis regimen other than 3 times weekly
* In ability to understand the English language and give informed consent for participation in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-11; Primary Completion 2011-02 (Actual); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Clearance of specific waste products from blood determined through subject blood and dialysate samples | 3 weeks

SECONDARY OUTCOMES:
Inflammation as determined by levels of specific inflammatory markers | 3 weeks
Red blood cell lifespan determined through a measurement of CO in the subject's breath | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nathan W. Levin, MD, Principal Investigator — Renal Research Institute; Peter Kotanko, MD, Study Director — Renal Research Institute
Locations (3):
- United States (3):
  - Irving Place Dialysis Center, New York, New York
  - Upper Manhattan Dialysis Center, New York, New York
  - Yorkville Dialysis Center, New York, New York

REFERENCES:
- [Derived] Rosales L, Thijssen S, Kruse A, Sipahioglu MH, Hirachan P, Raimann JG, Kuntsevich V, Carter M, Levin NW, Kotanko P. Inflammatory Response to Sorbent Hemodialysis. ASAIO J. 2015 Jul-Aug;61(4):463-7. doi: 10.1097/MAT.0000000000000212. PMID 25710773